CLINICAL TRIAL: NCT07157605
Title: Oncological Safety of Spleen Preservation in Left Pancreatectomy for Pancreatic Ductal Adenocarcinoma (SPLENDID): Study Protocol for a Prospective Observational International Multicenter Study
Brief Title: Oncological Safety of Spleen Preservation in Left Pancreatectomy for Pancreatic Ductal Adenocarcinoma (SPLENDID)
Acronym: SPLENDID
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, M.G. Besselink, Professor of Surgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2024.0713
Record Dates: First submitted 2025-04-02; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer Resectable; Pancreatectomy
Keywords: pancreatic adenocarcinoma; PDAC; left pancreatectomy; distal pancreatectomy; splenectomy; splenic hilum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to determine how often lymph node metastases occur in the splenic hilum and surrounding fat in patients with left-sided pancreatic cancer.

The main question the study aims to answer is:

Is spleen removal necessary in all cases, or is the risk of lymph node metastases in the fat around the spleen low enough to reconsider this standard practice?

Currently, spleen removal is part of the standard treatment for patients with left-sided pancreatic cancer to ensure that any potential lymph node metastases in the surrounding fat are also removed. However, the likelihood of metastases in this area is low, and spleen removal carries risks.

This study is a first step toward changing the treatment approach. If the findings show that metastases in the fat around the spleen are rare, the next step will be a randomized trial to further investigate whether spleen removal is necessary.

DETAILED DESCRIPTION:
Splenectomy is routinely performed during surgical resection of left-sided pancreatic ductal adenocarcinoma (PDAC) with the primary aim to facilitate adequate lymphadenectomy. However, asplenia is associated with several risks, including overwhelming post-splenectomy sepsis, and an increased risk of the development of cancer. Until several years ago, splenectomy was also routine practice in the surgical treatment of gastric cancer. Recently, several studies have shown that spleen-preservation in patients with gastric cancer is safe and therefore current guidelines advise against splenectomy. The rate of involved lymph nodes (LNs) in the splenic hilum (LN station 10) described in literature differs from 0 to 10% of patients. In these studies, the definition of the splenic hilum is often unclear and therefore these outcomes are difficult to interpret. Spleen-preservation in left-sided pancreatectomy for PDAC is currently not common practice in The Netherlands and goes against treatment guidelines. Two retrospective studies have suggested that spleenpreservation did not impair oncological outcomes and that postoperative complications occurred less after spleen preservation. However, these studies were retrospective, single-center and only included a very small number of patients and are therefore not providing enough evidence to change current practice. The SPLENDID-project focuses on evaluating the oncological safety of spleen-preservation in patients with left-sided PDAC. A prospective cohort study will be performed including all patients who undergo a left-sided pancreatectomy with splenectomy. The specimens will be transected at the precise level were spleen preservation (with resection of splenic vessels) would be performed (after removal of the specimen). Ratio of LN involvement will be collected for both specimen parts. Additionally, oncological patient outcomes, including survival, will be collected. When the pathological assessment confirms a <9% LN involvement rate in the perihilar space, the next step will be to assess spleen preservation in an international, multicenter randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive adult patients (≥ 18 years) who undergo an open or minimally invasive (i.e., robot-assisted or laparoscopic) left-sided pancreatectomy with concomitant splenectomy for primary resectable, borderline resectable, and locally advanced left-sided PDAC

Exclusion Criteria:

* Tumor involvement or abutment of the spleen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from hospitals performing pancreatic surgery
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node metastasis in spleen-part | 1 month

SECONDARY OUTCOMES:
Predictors for the occurrence of lymph node metastasis in the spleen-part | 1 month
  A regression analysis will be performed to determine the predictors for the lymph node metastasis in the spleen part
Overall and disease-free survival | 1 year, 2 years, 5 years
  Overall survival was defined as the time interval from surgery to death from any cause, and disease-free survival was defined as the time between surgery to either recurrence or death from any cause. 1-year, 2-year, and 5-year survival rates will be determined. Also the cause of death will be described.
Predictors for overall and disease-free survival | 1-year, 2-year, and 5-year
  A multivariable regression analysis will determine independent prognostic factors for overall and disease-free survival (including whether lymph node metastases in the spleen part are an independent prognostic factor).
Recurrence | 1 year, 2 years, 5 years
Recurrence-free survival | 1 year, 2 years, 5 years
  defined as the interval between surgery and recurrence, will be determined.
Lymph node metastasis (in pancreas-part and overall) | 1 month
  in pathological assessment
Identification of left gastroepiploic vessels in spleen-part | 1 month
  in pathological assessment
Identification of pancreatic tissue in spleen-part | 1 month
  in pathological assessment
Distance from transection plane to tumor | 1 month
  in pathological assessement
Tumor deposits | 1 month
  in pathological assessment
Radical (R0) resection rate | 1 month
  in pathological assessment
Histopathological diagnosis | 1 month
  in pathological assessment
Postoperative complications | 90 days
Length of hospital stay | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Jony van Hilst, MD, PhD, Principal Investigator — Amsterdam UMC, location University of Amsterdam, Department of Surgery, Amsterdam, The Netherlands; Marc G Besselink, MD, PhD, professor, Principal Investigator — Amsterdam UMC, location University of Amsterdam, Department of Surgery, Amsterdam, The Netherlands
Locations (10):
- BenQ Hospital, Nanjing, China
- Konstantopoulio General Hospital, Athens, Greece
- Padova University Hospital, Padua, Italy
- Kyushu University Hospital, Fukuoka, Japan
- Netherlands (3):
  - Amsterdam UMC, Amsterdam
  - OLVG Hospital, Amsterdam
  - Leiden University Medical Center, Leiden
- Oslo University Hospital, Oslo, Norway
- Dr. Peset University Hospital, Valencia, Spain
- Linköping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bruna CL, van Hilst J, Esposito A, Kleive D, Falconi M, Primrose JN, Korrel M, Bianchi D, Zerbi A, Kokkola A, Butturini G, Bjornsson B, Morone M, Casadei R, Marudanayagam R, Besselink MG, Abu Hilal M; European Consortium on Minimally Invasive Pancreatic Surgery (E-MIPS). The value of splenectomy during left-sided pancreatectomy for pancreatic ductal adenocarcinoma: predefined subanalysis in the DIPLOMA randomized trial. Br J Surg. 2024 Aug 30;111(9):znae236. doi: 10.1093/bjs/znae236. No abstract available. PMID 39287489
- See also: Dutch Pancreatic Cancer Group — https://dpcg.nl/studie/splendid-studie/
- See also: E-MIPS consortium (English) — https://www.e-mips.com/splendid